CLINICAL TRIAL: NCT06335953
Title: Demonstration of ALIGN: Aligning Medications With What Matters Most
Brief Title: ALIGN: Aligning Medications With What Matters Most (Demonstration)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00418404; U54AG063546 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Polypharmacy; Alzheimer's Disease and Related Dementias; Mild Cognitive Impairment
Keywords: Deprescribing
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention consists of the following:
  1. Mailing a deprescribing educational brochure to PLWD and care partners;
  2. PLWD and/or care partners will receive a single telehealth visit in which an embedded clinical pharmacist discusses the benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences;
  3. Pharmacist-primary care provider (PCP) communication in which the pharmacist provides tailored deprescribing recommendations designed to be useful and actionable for the PCP.
  Interventions: Behavioral: Pharmacist-led deprescribing intervention
- Delayed intervention (wait list control) (Active Comparator): The intervention consists of the following:
  1. Mailing a deprescribing educational brochure to PLWD and care partners;
  2. PLWD and/or care partners will receive a single telehealth visit in which an embedded clinical pharmacist discusses the benefits and harms of the patient's medications with the patient and care partner in the context of their goals and preferences;
  3. Pharmacist-primary care provider (PCP) communication in which the pharmacist provides tailored deprescribing recommendations designed to be useful and actionable for the PCP.
  Interventions: Behavioral: Pharmacist-led deprescribing intervention

INTERVENTIONS:
Behavioral: Pharmacist-led deprescribing intervention — The intervention consists of the following strategies: 1) Pharmacists will participate in a 20-minute webinar and receive a laminated tip sheet about the study; 2) Eligible patients and their care partners will receive a single deprescribing educational brochure by mail; 3) Patients and their care partners will have a single telemedicine visit in which the pharmacist will perform medication reconciliation and identify potential adverse effects and concerns related to medicines; 4) The pharmacist will send the PCP up to 3 deprescribing recommendations in the EHR using a standardized template; 5) With the PCP's approval, the pharmacist will call the patient or care partner to implement the deprescribing recommendations and document changes in the EHR.

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a pharmacist-led, primary care-based de-prescribing intervention for people living with dementia (PLWD) and the person's care partners.

The intervention consists of the following strategies: 1) a de-prescribing educational brochure designed to activate the patient and care partner; 2) a single telehealth visit in which an embedded clinical pharmacist discusses the benefits and harms of the patient's medications with the patient and care partner in the context of the person's goals and preferences; and 3) pharmacist-PCP communication in which the pharmacist provides tailored de-prescribing recommendations designed to be useful and actionable for the PCP.

The investigators will compare the intervention group with the waitlist control group to see if there is a difference in the primary outcome, the proportion of patients who deprescribe at least one medication by 3 months.

DETAILED DESCRIPTION:
PLWD have high rates of polypharmacy. This is due to the high degree of comorbid illnesses and challenging behavioral and psychological symptoms such as apathy and agitation. Guidelines written for individual conditions increase polypharmacy and potentially inappropriate medication (PIM) use, in which risks of medications outweigh benefits, or medications may not align with treatment goals. PIM in PLWD include anticholingerics, psychotropics and opioids, which are prescribed to PLWD in rates that far exceed use in the general older adult population, in spite of the association with harms such as falls, negative cognitive effects, cardiac conduction abnormalities, respiratory suppression and death. Polypharmacy and PIM use among PLWD is associated with adverse drug events, emergency department visits, hospitalizations, and treatment burden, suggesting that in some situations, "the cure may have become the disease."

The use of these and other medications requires nuanced decision-making to balance potential benefits and harms for PLWD. In keeping with principles of person-centered care, people should be on the medicines that will help achieve the persons goals, but not medicines that are likely to be harmful or unhelpful.

Deprescribing statins, antihypertensives, and psychotropic medications in older adults has been shown to be safe, and may lead to improved quality of life, reductions in falls, and improvements in cognitive and psychomotor function. Lessons from successful interventions include the need to target primary care clinicians and patients, and to target more than one class of medications. Most deprescribing interventions have occurred in hospitals, long-term care facilities, or home healthcare, not in primary care - typically the first point of contact with the health care system for PLWD. Few deprescribing studies have addressed care partners of PLWD, despite the enormous strain faced due to medication-related tasks and the person's specific informational and decisional needs and conflicts. These are gaps that the proposed research would address.

The investigator's previous research has shown that care partners want primary care providers (PCPs) to discuss medication-related goals of care as dementia progresses, and to acknowledge the tradeoffs implicit in using medications for symptom management in PLWD. But PCPs cite time pressure and lack of guidance of when and how to stop medications for PLWD as barriers to having these conversations. Pharmacists are ideally suited to help address these problems by providing evidence-based, individualized deprescribing recommendations without increasing demands on PCP time.

The clinical trial consists of the following strategies: 1) direct-to-consumer deprescribing educational materials designed to activate the care partner and PLWD; 2) telehealth visit in which a pharmacist discusses benefits and harms of the medications with the patient and care partner in the context of the person's goals and preferences; and 3) pharmacist-PCP communication in which the pharmacist provides tailored deprescribing recommendations that are actionable for the PCP. Pharmacists will receive a laminated tip sheet and participate in a 20-minute webinar. Decisions about discontinuation or continuation of medications will ultimately be made by the PCP and patient/care partner.

The trial is designed as a cluster-randomized trial with a delayed (waitlist) control where the unit of randomization will be the clinic. The investigators will enroll 280 patients with 140 per group (intervention group and waitlist control group). PLWD may enroll independently or together with a care partner. Care partners are not required to participate but may do so independently or with the PLWD if desired. Each participant will be in the study approximately 3 months (intervention period and additional follow-up).

This protocol employs a pragmatic design. The intervention is delivered by clinical pharmacists who are integrated in primary care clinics or practice through a centralized telemedicine model.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Diagnosis of dementia from International Classification of Diseases (ICD-10) visit codes or from the EHR problem list
* Five or more medications
* Only active patients, defined as having >1 visit to the primary care clinic within the past year will be included

Care partners:

* Family or other companions >21 years old who regularly help the patient manage medications.

Exclusion Criteria:

* As the pragmatic trial will be based on primary care, individuals residing in long-term care facilities or enrolled in hospice will be excluded.
* Participants must hear well enough to communicate by telephone in English.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 360 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-10-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who stop one or more medications | 3 months
  The primary outcome for the study will be the proportion of patients who stop ≥1 medication, assessed at 3 months. Discontinuation will be defined as a medication that is listed on the medication list at one time point and not listed at the subsequent time point.
  Discontinued medications will be measured using data obtained from the Electronic Health Record (EHR).

SECONDARY OUTCOMES:
Proportion of patients who start one or more new medications | 3 months
  The secondary outcome of the proportion of patients who start ≥1 medication will be assessed at 3 months. The start of a medication will be defined as a medication that is not listed on the medication list at one time point and listed at the subsequent time point.
  New medications started will be measured using data obtained from the EHR.
Proportion of patients who stop one or more potentially inappropriate medication (PIM) | 3 months
  The secondary outcome of the proportion of patients who stop ≥1 potentially inappropriate medication (PIM) will be assessed at 3 months. Discontinuation of a PIM will be defined as a PIM that is listed on the medication list at one time point and not listed at the subsequent time point.
  Discontinued PIM will be measured using data obtained from the EHR.
Total number of medications | Baseline and 3 months
  Total medication count will be measured using data obtained from the EHR.

OTHER OUTCOMES:
Shared decision-making as assessed by CollaboRATE | Immediately pre-pharmacist intervention, Immediately post-pharmacist intervention
  This is an exploratory, patient/care partner-reported outcome measure of shared decision-making. COLLABORATE uses a 9 point Likert scale that includes 3 questions. Score range 0-36. Higher scores represent better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Green, MD, MPH, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Community Physicians, Baltimore, Maryland, United States

REFERENCES:
- [Background] Alzheimer's Association. 2015 Alzheimer's disease facts and figures. Alzheimers Dement. 2015 Mar;11(3):332-84. doi: 10.1016/j.jalz.2015.02.003. PMID 25984581
- [Background] Davydow DS, Zivin K, Katon WJ, Pontone GM, Chwastiak L, Langa KM, Iwashyna TJ. Neuropsychiatric disorders and potentially preventable hospitalizations in a prospective cohort study of older Americans. J Gen Intern Med. 2014 Oct;29(10):1362-71. doi: 10.1007/s11606-014-2916-8. PMID 24939712
- [Background] Boyd CM, Darer J, Boult C, Fried LP, Boult L, Wu AW. Clinical practice guidelines and quality of care for older patients with multiple comorbid diseases: implications for pay for performance. JAMA. 2005 Aug 10;294(6):716-24. doi: 10.1001/jama.294.6.716. PMID 16091574
- [Background] Maust DT, Strominger J, Kim HM, Langa KM, Bynum JPW, Chang CH, Kales HC, Zivin K, Solway E, Marcus SC. Prevalence of Central Nervous System-Active Polypharmacy Among Older Adults With Dementia in the US. JAMA. 2021 Mar 9;325(10):952-961. doi: 10.1001/jama.2021.1195. PMID 33687462
- [Background] Carnahan RM, Lund BC, Perry PJ, Chrischilles EA. The concurrent use of anticholinergics and cholinesterase inhibitors: rare event or common practice? J Am Geriatr Soc. 2004 Dec;52(12):2082-7. doi: 10.1111/j.1532-5415.2004.52563.x. PMID 15571547
- [Background] Hill-Taylor B, Sketris I, Hayden J, Byrne S, O'Sullivan D, Christie R. Application of the STOPP/START criteria: a systematic review of the prevalence of potentially inappropriate prescribing in older adults, and evidence of clinical, humanistic and economic impact. J Clin Pharm Ther. 2013 Oct;38(5):360-72. doi: 10.1111/jcpt.12059. Epub 2013 Apr 2. PMID 23550814
- [Background] Castelino RL, Hilmer SN, Bajorek BV, Nishtala P, Chen TF. Drug Burden Index and potentially inappropriate medications in community-dwelling older people: the impact of Home Medicines Review. Drugs Aging. 2010 Feb 1;27(2):135-48. doi: 10.2165/11531560-000000000-00000. PMID 20104939
- [Background] Brown JD, Hutchison LC, Li C, Painter JT, Martin BC. Predictive Validity of the Beers and Screening Tool of Older Persons' Potentially Inappropriate Prescriptions (STOPP) Criteria to Detect Adverse Drug Events, Hospitalizations, and Emergency Department Visits in the United States. J Am Geriatr Soc. 2016 Jan;64(1):22-30. doi: 10.1111/jgs.13884. PMID 26782849
- [Background] Gray SL, Anderson ML, Dublin S, Hanlon JT, Hubbard R, Walker R, Yu O, Crane PK, Larson EB. Cumulative use of strong anticholinergics and incident dementia: a prospective cohort study. JAMA Intern Med. 2015 Mar;175(3):401-7. doi: 10.1001/jamainternmed.2014.7663. PMID 25621434
- [Background] Wimmer BC, Cross AJ, Jokanovic N, Wiese MD, George J, Johnell K, Diug B, Bell JS. Clinical Outcomes Associated with Medication Regimen Complexity in Older People: A Systematic Review. J Am Geriatr Soc. 2017 Apr;65(4):747-753. doi: 10.1111/jgs.14682. Epub 2016 Dec 19. PMID 27991653
- [Background] Page AT, Clifford RM, Potter K, Schwartz D, Etherton-Beer CD. The feasibility and effect of deprescribing in older adults on mortality and health: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Sep;82(3):583-623. doi: 10.1111/bcp.12975. Epub 2016 Jun 13. PMID 27077231
- [Background] Jansen J, Naganathan V, Carter SM, McLachlan AJ, Nickel B, Irwig L, Bonner C, Doust J, Colvin J, Heaney A, Turner R, McCaffery K. Too much medicine in older people? Deprescribing through shared decision making. BMJ. 2016 Jun 3;353:i2893. doi: 10.1136/bmj.i2893. No abstract available. PMID 27260319
- [Background] Scott IA, Hilmer SN, Reeve E, Potter K, Le Couteur D, Rigby D, Gnjidic D, Del Mar CB, Roughead EE, Page A, Jansen J, Martin JH. Reducing inappropriate polypharmacy: the process of deprescribing. JAMA Intern Med. 2015 May;175(5):827-34. doi: 10.1001/jamainternmed.2015.0324. PMID 25798731
- [Background] Kutner JS, Blatchford PJ, Taylor DH Jr, Ritchie CS, Bull JH, Fairclough DL, Hanson LC, LeBlanc TW, Samsa GP, Wolf S, Aziz NM, Currow DC, Ferrell B, Wagner-Johnston N, Zafar SY, Cleary JF, Dev S, Goode PS, Kamal AH, Kassner C, Kvale EA, McCallum JG, Ogunseitan AB, Pantilat SZ, Portenoy RK, Prince-Paul M, Sloan JA, Swetz KM, Von Gunten CF, Abernethy AP. Safety and benefit of discontinuing statin therapy in the setting of advanced, life-limiting illness: a randomized clinical trial. JAMA Intern Med. 2015 May;175(5):691-700. doi: 10.1001/jamainternmed.2015.0289. PMID 25798575
- [Background] Iyer S, Naganathan V, McLachlan AJ, Le Couteur DG. Medication withdrawal trials in people aged 65 years and older: a systematic review. Drugs Aging. 2008;25(12):1021-31. doi: 10.2165/0002512-200825120-00004. PMID 19021301
- [Background] van der Cammen TJ, Rajkumar C, Onder G, Sterke CS, Petrovic M. Drug cessation in complex older adults: time for action. Age Ageing. 2014 Jan;43(1):20-5. doi: 10.1093/ageing/aft166. Epub 2013 Nov 12. PMID 24222659
- [Background] Elliott RA, O'Callaghan C, Paul E, George J. Impact of an intervention to reduce medication regimen complexity for older hospital inpatients. Int J Clin Pharm. 2013 Apr;35(2):217-24. doi: 10.1007/s11096-012-9730-3. Epub 2012 Dec 5. PMID 23212732
- [Background] Sluggett JK, Hopkins RE, Chen EY, Ilomaki J, Corlis M, Van Emden J, Hogan M, Caporale T, Ooi CE, Hilmer SN, Bell JS. Impact of Medication Regimen Simplification on Medication Administration Times and Health Outcomes in Residential Aged Care: 12 Month Follow Up of the SIMPLER Randomized Controlled Trial. J Clin Med. 2020 Apr 8;9(4):1053. doi: 10.3390/jcm9041053. PMID 32276360
- [Background] Sheehan OC, Kharrazi H, Carl KJ, Leff B, Wolff JL, Roth DL, Gabbard J, Boyd CM. Helping Older Adults Improve Their Medication Experience (HOME) by Addressing Medication Regimen Complexity in Home Healthcare. Home Healthc Now. 2018 Jan/Feb;36(1):10-19. doi: 10.1097/NHH.0000000000000632. PMID 29298192
- [Background] Kerns JW, Winter JD, Winter KM, Kerns CC, Etz RS. Caregiver Perspectives About Using Antipsychotics and Other Medications for Symptoms of Dementia. Gerontologist. 2018 Mar 19;58(2):e35-e45. doi: 10.1093/geront/gnx042. PMID 28402533
- [Background] Green AR, Boyd CM, Gleason KS, Wright L, Kraus CR, Bedoy R, Sanchez B, Norton J, Sheehan OC, Wolff JL, Reeve E, Maciejewski ML, Weffald LA, Bayliss EA. Designing a Primary Care-Based Deprescribing Intervention for Patients with Dementia and Multiple Chronic Conditions: a Qualitative Study. J Gen Intern Med. 2020 Dec;35(12):3556-3563. doi: 10.1007/s11606-020-06063-y. Epub 2020 Jul 29. PMID 32728959
- [Background] Green AR, Lee P, Reeve E, Wolff JL, Chen CCG, Kruzan R, Boyd CM. Clinicians' Perspectives on Barriers and Enablers of Optimal Prescribing in Patients with Dementia and Coexisting Conditions. J Am Board Fam Med. 2019 May-Jun;32(3):383-391. doi: 10.3122/jabfm.2019.03.180335. PMID 31068402
- [Background] Reeve E, Bell JS, Hilmer SN. Barriers to Optimising Prescribing and Deprescribing in Older Adults with Dementia: A Narrative Review. Curr Clin Pharmacol. 2015;10(3):168-77. doi: 10.2174/157488471003150820150330. PMID 26338170